CLINICAL TRIAL: NCT05261386
Title: A Phase 2 Multicenter, Double-masked, Randomized, Vehicle-controlled, Parallel Study to Evaluate the Safety, Efficacy and Pharmacokinetics of CBT-008 in Patients With Meibomian Gland Dysfunction
Brief Title: Safety, Efficacy and Pharmacokinetics of CBT-008 in Patients With Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cloudbreak Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBT-CS-105
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2022-02

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Comparator: CBT-008 (Placebo Comparator): Vehicle
  Interventions: Drug: CBT-008
- Experimental: CBT-008 lower concentration (Experimental): lower concentration dose
  Interventions: Drug: CBT-008
- Experimental: CBT-008 higher concentration (Experimental): higher concentration dose
  Interventions: Drug: CBT-008

INTERVENTIONS:
Drug: CBT-008 — Treat MGD

SUMMARY:
Study Design

Structure: Multicenter, randomized, double-masked, vehicle-controlled, parallel group study Duration: 1 month of TID treatment Treatment Groups, Dosing, and Treatment Regimen Study Treatment: CBT-008 topical ophthalmic solution Control Treatment: CBT-008 vehicle

DETAILED DESCRIPTION:
Structure Multicenter, randomized, double-masked, vehicle-controlled, parallel group study.

Duration Stage 1: 1 month Stage 2: 1 day (1 dose)

Treatment Groups, Dosing, and Treatment Regimen

1. Study Treatment Stage 1: CBT-008 ophthalmic solution was administered as 1 drop OU TID Stage 2: CBT-008 ophthalmic solution was administered as 1 drop in the study eye
2. Control Treatment CBT-008 vehicle
3. Methods for Masking Study medication will be packaged in identical kits and will be labeled with medication kit numbers. The central randomization system will provide the site with a specific medication kit number for the patient corresponding to the treatment group assigned.
4. Instructions for Storage, Use, and Administration Study medication will be supplied as preservative free-unit dose containers, where 1 mL of CBT-008 ophthalmic solution will be aseptically filled into 3 mL Low Density Polyethylene (LDPE) ophthalmic dropper bottles. Study medication should be stored at room temperature in a secure area at clinical sites and dispensed only to patients enrolled into the clinical study. Patients will be instructed to store study medication in a cool place at room temperature at home. Study medication will be administered TID, one drop, to both eyes. First instillation of study medication on the first day will be applied by subject or care provider with site staff's observation for training and supervision. During the rest of the study treatment, patients will self-administer the medication TID for 1 month.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 inclusion criteria

* • Diagnosed with MGD in both eyes and meet the following:

  1. Ocular discomfort Score (ODS) ≥ 2 (No discomfort = 0, slight discomfort = 1, mild discomfort = 2, moderate discomfort = 3, severe discomfort = 4)
  2. Visual Analog Scale (VAS) level is 35-90% for at least 1 of the 7 categories
  3. Total Cornea staining grade ≥ 3 (NEI scheme with max score = 15)
  4. Total meibum quality score (MQS) is between 6-17 from the sum of the 6 lower eyelid central glands in at least one lower eyelid (0-3 scale with max total = 18).
  5. TBUT ≤ 5 s
  6. Schirmer I Test (anaesthetized) ≥ 5 mm/5 min in study eye
  7. BCVA LogMAR ≥ +0.7 in each eye

     * All patients of both genders ≥ 18 years
     * Willing to withhold the use of artificial tears and lubricants during the treatment phase;
     * Able to provide written informed consent and comply with study assessments for the full duration of the study.

Stage 2 inclusion criteria

1. Patients who completed the Stage 1 Exit Visit for at least 1 month or healthy volunteers
2. At least 18 years of age at time of consent and able to provide written informed consent

Exclusion Criteria:

Stage 1 exclusion criteria

* Uncontrolled systemic disease in the opinion of the Investigator

  * Active allergies with symptoms that may confound the data, active ocular infection requiring treatment, or ocular surface inflammatory disease unrelated to MGD or DED, including chalazion, inflamed pinguecula, and viral illness
  * History of ocular herpes disease in either eye
  * Incisional ocular surgery within 6 months or ocular laser surgery within 3 months
  * Use of topical treatment of the eye/eyelid with antibiotics, NSAIDS, or vasoconstrictors to treat MGD or DED within 14 days of screening; steroids, cyclosporin A or lifitegrast within 28 days of screening
  * Current or anticipated use of other topical ophthalmic medications in the study eye. (Patients must have discontinued the use of ophthalmic medications in the study eye for at least 2 weeks prior to the screening visit, the use of diagnostic medications as part of the eye exam prior to screening and artificial tears is allowed.)
  * Anticipated wearing of contact lenses during any portion of the study. (Patients, who wear soft contact lenses should discontinue wearing them at least 3 days prior to screening visit. Patients wearing rigid gas permeable or hard contact lenses should discontinue wearing them at least 3 weeks prior to screening visit.)
  * Active rosacea involving the eyelids within 60 days of screening
  * Current enrollment in an investigational drug or device study or participation in such a study within 30 days prior to entry into this study
  * Any condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
  * Female patients who are pregnant, nursing, or planning a pregnancy during the study Stage 2 exclusion criteria

    1. Females who were pregnant or nursing
    2. Current enrollment in an investigational drug or device study or participation in such a study within 30 days prior to entry into this study
    3. Previously randomized in the CBT-CS102 clinical trial and dosed with CBT-006

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bing Leng, MD, Study Director — ADS Therapeutics, LLC
Locations (1):
- David Research Wirta, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT-008 Vehicle: Vehicle CBT-008: ophthalmic solution
- Experimental: Lower Concentration CBT-008: lower concentration CBT-008 ophthalmic solution
- Experimental: Higher Concentration CBT-008 CBT-008: Higher concentration CBT-008 ophthalmic solution. CBT-008
Period: Overall Study
Arm/Group | CBT-008 Vehicle | Experimental: Lower Concentration CBT-008 | Experimental: Higher Concentration CBT-008 CBT-008
Started | 32 | 31 | 32
Completed | 32 | 30 | 32
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CBT-008 Lower Concentration Ophthalmic Solution: lower concentration dose
  CBT-008: ophthalmic solution
- CBT-008 Higher Concentration Ophthalmic Solution: higher concentration dose
  CBT-008: ophthalmic solution
- Total: Total of all reporting groups
Arm/Group | CBT-008 Vehicle | CBT-008 Lower Concentration Ophthalmic Solution | CBT-008 Higher Concentration Ophthalmic Solution | Total
Number analyzed (Participants) | 32 | 31 | 32 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 19 | 19 | 61
  >=65 years | 9 | 12 | 13 | 34
Age, Continuous [Median (Standard Deviation); unit: years] | 56.5 (15.67) | 61.5 (10.75) | 62.6 (13.80) | 60.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 23 | 65
  Male | 7 | 14 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 4 | 20
  Not Hispanic or Latino | 24 | 23 | 28 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 5 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 6 | 17
  White | 19 | 20 | 19 | 58
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 32 | 95
Intraocular Pressure of study eye related to safety [Mean (Standard Deviation); unit: mmHg] | 15.844 (2.9415) | 16.371 (2.1015) | 16.078 (2.3352) | 16.098 (0,2156)

OUTCOME MEASURES:

1. Primary Outcome: IOP Related to Safety
Description: Intraocular Pressure for study eye
Time Frame: 4 weeks
Population: Safety Population Study eye
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- CBT-008 Ophthalmic Solution: Vehicle
  CBT-008: ophthalmic solution
- CBT-008 Lower Concentration: CBT-008 ophthalmic solution lower concentration dose
- CBT-008 Higher Concentration: higher concentration dose CBT-008 ophthalmic solution
Arm/Group | CBT-008 Ophthalmic Solution | CBT-008 Lower Concentration | CBT-008 Higher Concentration
Number analyzed (Participants) | 32 | 31 | 32
mmHg | 15.906 (3.0860) | 16.452 (2.6999) | 16.469 (2.2823)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Vehicle: One drop in the study administered three times daily (TID)
  Vehicle: One drop in the study administered three times daily (TID) for 4 weeks
- CBT-008 Ophthalmic Solution Single Dose; CBT-008 Ophthalmic Solution Multi-dose: One drop in the study administered three times daily (TID)
  CBT-008: One drop in the study administered three times daily (TID) for 4 weeks
Arm/Group | Vehicle | CBT-008 Ophthalmic Solution Single Dose | CBT-008 Ophthalmic Solution Multi-dose
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 3/32 | 5/31 | 8/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=32) | CBT-008 Ophthalmic Solution Single Dose (N=31) | CBT-008 Ophthalmic Solution Multi-dose (N=32)
Non-ocular TEAEs (General disorders) | 0 (0) | 1 | 2
Ocular TEAEs (Eye disorders) | 3 (3) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT05261386/Prot_SAP_ICF_000.pdf